CLINICAL TRIAL: NCT02927821
Title: Improving Outcome for Family Caregivers of Older Adults With Complex Conditions: The Adult Day Plus (ADS Plus) Program
Acronym: ADS Plus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Minnesota (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00112546; 1R01AG049692-01 (NIH)
Record Dates: First submitted 2016-08-19; First posted 2016-10-07 (Estimated); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Stress
Keywords: Adult Day Care Centers; Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ADS Plus (Experimental): Families in settings assigned to intervention will receive Adult Day Services (ADS) as usual in addition to ADS Plus. ADS Plus has 5 key components: care management, referral/linkage; disease education; counseling/emotional support/stress reduction, and care skills managing daily challenges and behavioral disturbances. The intervention begins with 2 face-to-face sessions with the site interventionist to conduct a needs assessment to identify concerns and needs and develop an agreed upon care plan. The interventionist then meets with caregivers face-to-face at convenient times to implement the care plan, every other week for the first 3 months, and then for monthly reassessments for newly emerging care concerns thereafter. Contact occurs about a minimum of 1 hour per month over 12 months.
  Interventions: Behavioral: ADS Plus
- ADS Usual Care (No Intervention): Caregivers in the 15 sites assigned to serve as the usual care control group will receive Adult Day Services (ADS) as usual. Near completion of the study (project year 05), control group sites will have the option of receiving training in ADS Plus for their setting.

INTERVENTIONS:
Behavioral: ADS Plus — Contact occurs at a minimum for about 1 hour per month over 12 months (face-to-face/ telephone). Targeted education materials concerning clients' conditions and related matters are shared via email or traditional mail. The goal of each contact is to provide ongoing emotional support, situational counseling, education about importance of taking care of self, referrals/linkages and skills (e.g., stress reduction, behavioral management, how to talk with doctors). The care planning process is collaborative and flexible, reflecting CG fluctuating needs
  Other Names: Adult Day Services Plus; ADS+
  Arms: ADS Plus

SUMMARY:
Over 15 million family caregivers provide more than 85% of long-term care to older adults with Alzheimer's Disease and Related Disorders. Caregivers typically assume care responsibilities without training or support and may in turn experience multiple health risks including depression. Providing evidence-based caregiver supportive programs on a wide scale basis is identified by the National Alzheimer's Plan Act as a national priority. One approach is to augment existing community-based services for older adults with a caregiver evidence-based program. Adult day service (ADS) is one such growing and critical community-based option for older adults with Alzheimer's Disease and related disorders but which does not systematically address common caregiver challenges or burdens using evidence-based programs. The purpose of the study is to: 1) evaluate the effectiveness of Adult Day Services (ADS) Plus to improve caregiver well-being and reduce depressive symptoms compared to routine ADS use at 6 months; and 2) evaluate long-term maintenance effects of ADS Plus at 12 months on caregiver well-being and depressive symptoms. ADS Plus consists of 5 key components: care management, referral/linkage, education about dementia, situational counseling/emotional support/stress reduction techniques, and skills to manage behavioral symptoms (e.g., rejection of care, agitation, aggression). Based on care challenges identified by family caregivers, an "ADS Plus Prescription" is provided, a written document detailing easy-to-use strategies to address specified care challenges and caregivers are trained in their use. The proposed study will employ a practical trial design to assess the effectiveness and uptake of ADS Plus on a large scale. Thirty ADS programs throughout the U.S. varying in geographic location and staffing levels will be involved. A total of 300 diverse caregivers (150 in 15 ADS Plus sites; 150 in 15 ADS usual care sites) will be enrolled.

DETAILED DESCRIPTION:
Family caregivers (CGs) provide 85% or more of the long-term care needs of older adults including coordination, care transitions, hands-on assistance with daily care, health-related services (e.g., wound care, medication management), financial support, monitoring on-site or long-distance, managing challenging behaviors, and preserving quality of life. As conditions worsen, CGs assume more extensive care responsibilities that can be time consuming, physically demanding, and emotionally depleting. Although positive aspects of caregiving are documented, on-going caregiving can be a source of chronic stress resulting in poor health, lost income, psychological distress, and for those most distressed, increased risk of mortality.

CGs typically provide care without formal support, have significant unmet needs, and limited access to the knowledge and skills needed to care for older adults with complex conditions. To date, most tested CG interventions have: a) focused on one disease state (e.g., dementia); b) delivered interventions outside existing service settings/payment structures; c) required extensive training of interventionists, d) had less reach to a mix of CGs/older persons; e) required retooling of the intervention to enhance its implementation potential in real world settings; and f) not been translated for delivery in community-settings nor sustained. The study potentially overcomes these shortcomings by embedding an evidence-based approach in a service and payment structure (adult day services [ADS]), addressing core needs of diverse CGs of older adults with a mix of conditions, and evaluating outcomes of high relevance to CGs (well-being, depression), older adults (behavioral symptoms), ADS (more days spent in ADS) and society (reduction of nursing home placement).

Adult day services are a growing and important long-term care option. ADS is an important community-based long-term care option for CGs and older adults with complex conditions requiring daily assistance. ADS provides out-of-home, supervised, group services with the goals of improving mood, well-being, and quality of life and enabling clients to remain at home for as long as possible. ADS also aims to provide CGs "respite" from day-to-day care responsibilities and is available during "normal business hours," although some offer flexible hours to meet the needs of working CGs. While some provide support groups and educational opportunities, these activities are not consistently provided, systematically integrated into routine practice, or evidence-based. Similarly, while some care planning may occur at the time of client enrollment or annually, structured, consistent contacts with CGs using standardized assessments and evidence-based approaches are not typically offered. The intervention being evaluated, ADS Plus, is evidence-driven, embedded in ADS work flow, and systematically addresses unmet CG needs that may boost ADS benefits for both CGs and older adult clients.

The primary study aims are to: 1) evaluate the effectiveness of ADS Plus to improve CG well-being and reduce depressive symptoms compared to routine ADS use at 6 months; and 2) evaluate long-term maintenance effects of ADS Plus at 12 months on CG well-being and depressive symptoms.

Additional study aims will: 3) evaluate whether CGs using ADS Plus are more likely to maintain relatives in ADS and less likely to place them in residential settings compared to those in routine ADS over 12 months; 4) estimate ADS Plus costs and assess whether it results in net financial benefits when compared to usual ADS at 6 and 12 months; 5) evaluate the effects of ADS Plus on client behaviors and CG efficacy and upset managing symptoms; and 6) evaluate theoretically-derived ( Reach Effectiveness Adoption Implementation Maintenance (RE-AIM) framework, Stress Process Model) mediational pathways of treatment change including CG acceptance and staff adoption of ADS Plus over 12 months.

Overview of research design. The investigators propose a two group cluster randomized trial using re-randomization and mixed methods to combine effectiveness and implementation questions to enhance the yield of this translational study.

This hybrid (also called a practical or embedded trial) will involve 30 ADS sites located across the U.S. that will be randomized into two groups: 15 ADS programs will serve as treatment sites and provide ADS services as usual and the ADS Plus intervention; 15 ADS programs will serve as the control condition and will provide ADS as usual. Prior to randomization, the investigators will carefully examine sites on important variables such as size or capacity, location (urban, suburban, rural), percent of participants with a dementia diagnosis, staff to client ratio, ownership structure, and how long each center has been operating. The investigators will then implement re-randomization techniques to ensure optimal balance between ADS Plus and control sites on these site-level factors. Each of 30 sites will enroll 15-23 CGs in the study, with the expectation that an average of 10 per site will be retained at 6 months (43% attrition projected based on ADS Plus pilot and other CG trials). This will yield a total of 300 retained participants (150 CGs in ADS Plus sites; 150 in ADS usual care sites) over a 2 year recruitment period. In accordance with the translational focus, the inclusion criteria are purposely broad to reflect the real world case mix of CGs using ADS such that any CG with an older relative (>60 years) upon initial intake and enrollment in a participating ADS will be eligible for study inclusion. Each of 30 ADS sites will designate a staff member to serve as research liaison for that site and participate in 4 hours of paid training (via webinar). Research liaisons will be responsible for informing CGs (at initial intake) of the study using Johns Hopkins University (JHU) approved Institutional Review Board (IRB) scripts, recruitment letters and flyers. The Research liaisons will provide a packet of study materials that will contain a copy of the consent form, study flyer, study letter, consent to contact sheet. CGs expressing study interest will sign an IRB approved form to agree to be contacted by study staff. Caregivers will receive a telephone call from a JHU research interviewer. The interviewer will explain study procedures, review the consent form that the caregiver has been provided in the packet. If the caregiver is interested the staff will obtain verbal assent and instruct the caregiver to sign the consent form with the date and time. If the CG is eligible and has signed the consent and provided verbal assent a 45 minute baseline interview will be conducted either immediately or at a time convenient for the CG yet within 1 week of screening. The consent form will then be returned to the ADS site and scanned or faxed to JHU study staff. In previous trials, the investigators found CGs can attend to an hour by telephone.

The 15 ADS Plus sites will also designate a site interventionist and a backup interventionist who will participate in up to one week of training (via webinar, on-line lectures) in ADS Plus protocols. For those in ADS Plus sites, once the baseline interview is completed the JHU project director will inform the site interventionist to contact that CG and begin ADS Plus (to occur within 10 days from baseline interview). All CGs (treatment/control) will be interviewed via telephone by JHU research staff at 3 months (interim check-in for retention and collect data on key CG outcomes), 6 months (main trial outcome for CG benefits), and 12 months (long-term outcomes for older adult clients and CG). To evaluate implementation processes, interviewers at the University of Minnesota (UoM) will administer a brief checklist at 6 and 12-months to CGs (n=150) from the 15 ADS Plus sites and to the 15 ADS Plus interventionists. Additionally, at 12-months the 15 ADS Plus interventionists will be surveyed using semi-structured interviews by telephone to collect detailed process data on treatment fidelity. These interviews will ascertain challenges and successes of administering ADS Plus to identify areas to refine prior to ADS Plus dissemination in the final phases of the proposed project. Also, at the conclusion of the randomized control trial (RCT), 20 of 150 CGs from the 15 ADS Plus sites will be purposively sampled (based on CG relationship, gender, race/ethnicity, and cognitive impairment of client) to participate in a post-RCT qualitative interview. A semi-structured telephone interview conducted by UoM interviewers will explore how ADS Plus helped them (or not) and perceptions concerning effects of the intervention for clients.

Description of ADS Plus. Theoretical Framework - ADS Plus draws upon the Pearlin et al., stress process model and its iteration in the NIH REACH trials. These models suggest that factors such as care needs of older adults, behavioral symptoms, and/or CG health serve as primary stressors for CGs. CGs evaluate whether external demands pose potential threats to the older adult and/or themselves, and if so, whether they have sufficient coping mechanisms. If CGs perceive external demands as threatening and their coping resources as inadequate, they experience burden. The appraisal of stress is assumed to contribute to negative emotional, physiological, and behavioral responses that place CGs at risk for poor health, diminished wellbeing and depression.

Delivery Characteristics - Families in settings assigned to intervention will receive ADS as usual in addition to ADS Plus. ADS Plus consists of 5 key components: care management, referral/linkage; disease education; counseling/emotional support/stress reduction, and care skills managing daily challenges and behavioral disturbances (e.g., rejection of care). Each component is tailored to CGs' unmet needs and care context. The intervention begins with two face-to-face sessions with the appointed site interventionist to conduct a systematic needs assessment from which to identify concerns and needs and develop an agreed upon care plan. The interventionist then meets with CGs face-to-face at convenient times (e.g., when relative is brought to or picked up at ADS) to implement the care plan, every other week for the first 3 months, and then for monthly reassessments for newly emerging care concerns thereafter. Contact occurs at a minimum for about 1 hour per month over 12 months (face-to-face/ telephone). Targeted education materials concerning clients' conditions and related matters are shared via email or traditional mail. The goal of each contact is to provide ongoing emotional support, situational counseling, education about importance of taking care of self, referrals/linkages and skills (e.g., stress reduction, behavioral management, how to talk with doctors). The care planning process is collaborative and flexible, reflecting CG fluctuating needs Usual care control group: CGs in the 15 sites assigned to serve as the usual care control group will receive ADS as usual. As the study intent is to demonstrate the added value of ADS Plus, comparing it to ADS (usual care) is appropriate and reflects the translational purpose of the proposed study. Near completion of the study (project year 05), control group sites will have the option of receiving training in ADS Plus for their setting. As CGs in control sites would have completed the study prior to this training, it may benefit these sites and their future clients/families but not those enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

Caregivers are eligible to participate at time of intake at an Adult Day Service (ADS) if they:

* are initially enrolling their relative in one of the 30 participating ADS sites
* expect to use ADS for a minimum of 1 week for 6 months
* have primary responsibility for care of the ADS client
* speak English
* provided > 8 hours of assistance to client in past week
* have a telephone and are willing to participate in 4 telephone interviews (baseline, 3 month check-in; 6 and 12 month follow-ups)
* are 21 years of age or older (male or female).

Exclusion Criteria:

caregivers and older adult clients are not eligible if:

* they plan to move from the area within 6 months
* either caregiver or client has been hospitalized >3 times in past year
* either caregiver or client is in active treatment for a terminal illness or are in hospice
* caregiver is involved in other caregiver support services/trials.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2016-10; Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Improve Caregiver Well-being as assessed by the Perceived Change Scale | from baseline to 6 months
  Caregiver Well-being will be measured using Perceived Change Scale. This is a 13-item scaled scored on a 5-point Likert scale with 1 = gotten much worse to 5 = improved a lot with higher scores indicating better well-being.
Improve Caregiver Well-being as assessed by the Perceived Change Scale | from baseline to 12 months
  Caregiver Well-being will be measured using Perceived Change Scale. This is a 13-item scaled scored on a 5-point Likert scale with 1 = gotten much worse to 5 = improved a lot with higher scores indicating better well-being.
Decrease Depressive Symptoms in Caregivers as assessed by Center for Epidemiological Studies Depression Scale (CES-D). | from baseline to 6 months
  Caregiver depressive symptoms will be measured using the Center for Epidemiological Studies Depression Scale (CES-D). The CES-D is a 20 item scale, scored 0 to 3 for each item. Zero means rarely or none of the time and 3 means most or all of the time. Lower scores indicate less depressive symptoms.
Decrease Depressive Symptoms in Caregivers as assessed by Center for Epidemiological Studies Depression Scale (CES-D). | from baseline to 12 months
  Caregiver depressive symptoms will be measured using the Center for Epidemiological Studies Depression Scale (CES-D). The CES-D is a 20 item scale, scored 0 to 3 for each item. Zero means rarely or none of the time and 3 means most or all of the time. Lower scores indicate less depressive symptoms.

SECONDARY OUTCOMES:
Cost Analysis of Intervention as assessed by the Resource Utilization in Dementia (RUD) | baseline to 6 months
  Cost will be computed using the Resource Utilization in Dementia (RUD). The RUD scale assess use of social services, frequency and duration of hospitalizations, contact with health care professionals, time spent caring for the person with dementia, missed word and medication use.
Cost Analysis of Intervention as assessed by the Service Utilization and Resources Survey (SURF) | Baseline to 6 months
  Cost will be computed using the Service Utilization and Resources Survey (SURF). This survey asks about healthcare service use and time spent with care.
Improve Caregiver Well-being as reported on the Neuropsychological Inventory Questionnaire (NPI-Q) caregiver distress questions. | from baseline to 6 months
  Caregiver well-being will be measured using Caregiver stress as reported on the Neuropsychological Inventory Questionnaire (NPI-Q). The NPI-Q is a 12 item scale where caregiver distress is scored on a 6 point Likert Scale with zero equal to not at all distressing to 5 meaning extreme or very severe distress. Higher Scores indicate more distress.
Improve Caregiver Well-being as reported on the Neuropsychological Inventory Questionnaire (NPI-Q) caregiver distress questions. | from baseline to 12 months
  Caregiver well-being will be measured using Caregiver stress as reported on the Neuropsychological Inventory Questionnaire (NPI-Q). The NPI-Q is a 12 item scale where caregiver distress is scored on a 6 point Likert Scale with zero equal to not at all distressing to 5 meaning extreme or very severe distress. Higher Scores indicate more distress.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Gitlin, PhD, Principal Investigator — Johns Hopkins University; Joseph Gaugler, PhD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - Johns Hopkins, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gitlin LN, Reever K, Dennis MP, Mathieu E, Hauck WW. Enhancing quality of life of families who use adult day services: Short- and long-term effects of the adult day services plus program. Gerontologist. 2006 Oct;46(5):630-9. doi: 10.1093/geront/46.5.630. PMID 17050754
- [Derived] Gitlin LN, Marx KB, Roth DL, Anderson K, Dabelko-Schoeny H, Scerpella D, Parker LJ, Koeuth S, Gaugler JE. Fidelity matters: implementing ADS Plus, an evidence-based program, in multiple adult day service sites. Innov Aging. 2025 Jul 1;9(8):igaf074. doi: 10.1093/geroni/igaf074. eCollection 2025 Aug. PMID 40979469
- [Derived] Cotton QD, Bailey D, Albers E, Ingvalson S, Bloomquist E, Marx K, Anderson K, Dabelko-Schoeny H, Parker L, Gitlin LN, Gaugler JE. Understanding the implementation process of the Adult Day Services Plus program. BMC Geriatr. 2025 Feb 13;25(1):95. doi: 10.1186/s12877-025-05757-4. PMID 39948465
- [Derived] Gitlin LN, Roth DL, Marx K, Parker LJ, Koeuth S, Dabelko-Schoeny H, Anderson K, Gaugler JE. Embedding Caregiver Support Within Adult Day Services: Outcomes of a Multisite Trial. Gerontologist. 2024 Apr 1;64(4):gnad107. doi: 10.1093/geront/gnad107. PMID 37549428
- [Derived] Parker LJ, Marx KA, Nkimbeng M, Johnson E, Koeuth S, Gaugler JE, Gitlin LN. It's More Than Language: Cultural Adaptation of a Proven Dementia Care Intervention for Hispanic/Latino Caregivers. Gerontologist. 2023 Mar 21;63(3):558-567. doi: 10.1093/geront/gnac120. PMID 35951488
- [Derived] Gitlin LN, Marx K, Scerpella D, Dabelko-Schoeny H, Anderson KA, Huang J, Pizzi L, Jutkowitz E, Roth DL, Gaugler JE. Embedding caregiver support in community-based services for older adults: A multi-site randomized trial to test the Adult Day Service Plus Program (ADS Plus). Contemp Clin Trials. 2019 Aug;83:97-108. doi: 10.1016/j.cct.2019.06.010. Epub 2019 Jun 22. PMID 31238172